CLINICAL TRIAL: NCT01421758
Title: Using Facebook to Increase Social Support for Physical Activity: The INSHAPE Study
Brief Title: Testing the Efficacy of an Online Social Network Intervention to Increase Social Support for Physical Activity
Acronym: INSHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-1122
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2011-08

CONDITIONS: Cardiovascular Disease; Cancer; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Obesity | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- online social network (Experimental)
  Interventions: Behavioral: online social network enrollment plus education and self monitoring
- web education control (Active Comparator)
  Interventions: Behavioral: Web education control

INTERVENTIONS:
Behavioral: online social network enrollment plus education and self monitoring — Participants are enrolled in an online social network designed to increase social support for physical activity and will self monitor physical activity and receive educational materials at a dedicated study website.
  Arms: online social network
Behavioral: Web education control — Participants will receive access to a dedicated study website where they can view educational materials related to physical activity
  Arms: web education control

SUMMARY:
This study was designed to determine whether participation in an online social network intervention increases perceived social support for physical activity versus a minimal education control group by conducting a randomized controlled trial with 140 female undergraduate students. The investigators hypothesize that participants in the physical activity centered online social network intervention group will have greater increases in perceived social support for physical activity compared to minimal web based physical activity education controls.

ELIGIBILITY:
Inclusion Criteria:

* female
* under the age of 25
* currently enrolled full time or part time student at the University of North Carolina at Chapel Hill
* classified as an undergraduate
* answers no to all questions on an exercise risk factor questionnaire (PAR-Q) or is cleared in writing by a physician to participate in an independent exercise program
* a score of less than 3 on the SCOFF eating disorders questionnaire
* less than 30 minutes per day of self reported moderate or vigorous physical activity
* regular Facebook use as defined by self reported owning of an account and use of at least 30 minutes per day
* willing to provide informed consent
* willing to participate in the intervention
* literate in the English language.

Ages: 17 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mean perceived social support for physical activity scores on the Peer/Friend Support for Healthy Eating and Physical Activity Scale. | 10 weeks
  The primary outcome measure is the mean score of a 19 item, 7 point scale that measures the frequency of social support interactions over the previous 6 weeks.

SECONDARY OUTCOMES:
Physical activity in kilocalories on the Paffenbarger Physical Activity Questionnaire/College Alumnus Questionnaire | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David N Cavallo, MPH, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Cavallo DN, Tate DF, Ries AV, Brown JD, DeVellis RF, Ammerman AS. A social media-based physical activity intervention: a randomized controlled trial. Am J Prev Med. 2012 Nov;43(5):527-32. doi: 10.1016/j.amepre.2012.07.019. PMID 23079176